CLINICAL TRIAL: NCT02520609
Title: Dynamic Post-Prandial Metabolism in Patients With Non-Alcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150174; 15-DK-0174
Record Dates: First submitted 2015-08-08; First posted 2015-08-13 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-07-03

CONDITIONS: Liver Disease; Fatty Liver
Keywords: Metabolomics; Non-Alcoholic Steatohepatitis; Non-Alcoholic Fatty Liver Disease; Energy Expenditure; Natural History
MeSH Terms: conditions — Liver Diseases; Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Healthy volunteers
- Patients with metabolic syndrome without NAFLD: Patients with metabolic syndrome without NAFLD
- Patients with NAFLD: Patients with NAFLD

SUMMARY:
Background:

Metabolism refers to the many chemical pathways by which various compounds, including food, are processed and used in the body. People with non-alcoholic fatty liver disease (NAFLD) have too much fat in their liver cells, but what causes it is unclear. One explanation is that people with NAFLD process food and metabolize it differently than people without NAFLD. Researchers want to compare how food is metabolized in people with and without NAFLD.

Objective:

To better understand how food intake influences the development and progression of NAFLD.

Eligibility:

People ages 18 and older with NAFLD or with a non-NAFLD metabolic syndrome

Healthy volunteers ages 18 and older

Design:

Participants will be screened with medical history, surveys, physical exam, and blood tests. This will have ultrasound of the abdomen. This uses sound waves to image internal organs.

Participants will stay at the Clinical Center for 2 nights.

They will fast he first night.

On the second day they will:

Have their metabolism monitored in a metabolism research room for 24 hours

Have a catheter inserted into an arm vein for several blood tests

Drink an Ensure Plus for breakfast

Have solid meals for lunch and dinner

Have several urine tests.

The final morning, they will:

Have more blood tests.

Have a DXA test to measure the fat in the body. They will lie on their backs for 15-25 minutes while an x-ray machine is positioned over areas of the body.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common hepatic disorder in the Western world and is a leading cause of liver-related morbidity and mortality. Excessive caloric intake and specific nutritional components have been implicated in its pathogenesis, but the complex metabolic pathways linking nutrient consumption with hepatic fat accumulation have not yet been fully elucidated. Analysis of pathophysiology and the search for biomarkers in NAFLD has largely focused on fasting samples; the dynamic response to a caloric load has not been interrogated, beyond glucose tolerance testing. Metabolomics is a novel high-throughput technique, allowing for simultaneous detection of hundreds to thousands of metabolites, and the evaluation of their interconnectivity and causal relationships. We propose a pilot study to investigate the metabolic response of patients with NAFLD to a standardized food challenge, by applying a metabolomics-based dynamic approach. In this study we will recruit up to 50 patients with NAFLD and compare them to 12 controls with metabolic syndrome without NAFLD, and 12 healthy controls. Following an overnight fast, subjects will be situated in a metabolic chamber for continuous measurement of metabolic rates and will be given a liquid mixed meal containing approximately 30% of daily caloric requirement over a period of 15 minutes. The energy expenditure (EE) and respiratory quotient (RQ), reflecting preference for carbohydrate or fat oxidation, will be measured at 1-minute resolution. Blood will be drawn at baseline, and at 30 min, 1, 2, 4 and 24 hours after ingestion. Plasma will be separated and stored in -80 (Infinite)C. Following completion of recruitment, stored samples will be analyzed at the NCI Laboratory of Metabolism by LC/MS and GC/MS, metabolites of interest identified, and individual metabolites quantitated and normalized to their pre-prandial level. Study results will hopefully identify novel metabolic markers of disease, and uncover altered signaling pathways unique to NAFLD that are activated primarily under fed state conditions.

ELIGIBILITY:
* INCLUSION CRITERIA:

For the entire cohort:

* Male or female aged > 18 years
* Ability to provide informed consent

For group 1 subjects (NAFLD)

* Biopsy-proven NAFLD within 2 years prior to screening, OR
* The presence of at least two of the following criteria:
* Suggestion of liver fat by an imaging study (ultrasound, CT scan, MRI or MR spectroscopy) performed in the 6 months prior to screening
* Elevated aminotransferase levels (ALT > 31 U/L for men or > 19 U/L for women, or AST > 30 U/L) on at least two occasions in the 6 months preceding enrollment.
* Presence of the metabolic syndrome, defined according to the modified AHA/NCEP criteria as the presence of at least three of:

  i. Abdominal obesity, defined as waist circumference > 102 cm for men or > 88 cm for women

ii. Elevated triglycerides (> 150 mg/dL) or the use of medication to lower triglycerides

iii. Reduced HDL cholesterol (< 40 mg/DL for men or < 50 mg/dL for women)

iv. Elevated blood pressure (> 135/80 mmHg) or use of medication for hypertension

v. Elevated fasting glucose levels (> 100 mg/dL) or use of anti-diabetic medication

For the purpose of inclusion, the presence of overt diabetes mellitus type 2 will be considered equivalent to the presence of the metabolic syndrome, even if the other criteria are absent.

For group 2 subjects (non-NAFLD metabolic syndrome):

* Evidence of metabolic syndrome
* Normal transaminases (ALT less than or equal to 31 U/L for men or less than or equal to 19 U/L for women, or AST less than or equal to 30 U/L) at screening
* Absence of liver fat by imaging or liver biopsy within 6 months of screening

For group 3 subjects (healthy volunteers):

* No history of known liver disease
* Not on any regular systemic medications (with the exception of oral contraceptives)
* BMI <= 25 kg/m2
* Non diabetic
* Normal transaminases and fasting glucose (<95 mg/dL)

EXCLUSION CRITERIA:

1. Concomitant liver disease such as autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson s disease, alpha-1 antitrypsin deficiency
2. Chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV). Patients who were treated successfully for HCV and achieved sustained virological response can be eligible for enrollment > 18 months after treatment cessation. Patients receiving antiviral therapy are ineligible.
3. Estimated average alcohol consumption > 30 g/d for men or > 20 g/d for women in the 6 months prior to enrollment, or binge-drinking behavior .
4. Gain or loss of > 10% body weight within the 6 months prior to enrollment.
5. Decompensated liver cirrhosis, defined as a past or present occurrence of a decompensation event (variceal bleeding, ascites, spontaneous bacterial peritonitis, encephalopathy or hepatocellular carcinoma or by albumin < 3 g/dl, PT > 3 seconds above the upper limit of the norm, platelet count < 70,000 or total bilirubin > 2 mg/dL (in the absence of Gilbert s syndrome).
6. Pregnancy or lactation
7. Treatment with medications known to cause fatty liver disease such as atypical neuroleptics, tetracycline, methotrexate or tamoxifen
8. Disorders interfering with substrate absorption such as gastric bypass surgery, malabsorption disorders, use of orlistat or bile acid sequestrants, or extensive small bowel resection.
9. Diabetic patients requiring insulin treatment
10. Lactose intolerance or allergy to Ensure or one or more of its components
11. Hyper/hypothyroidism
12. Inability to remain sedentary for 4 hours, or to remain for 26-30 hours in the metabolic chamber
13. Inability to obtain vascular access for the required blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Metabolomics readout | One point measure
  Plasma metabolomic Readout

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rotman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0174.html